CLINICAL TRIAL: NCT01955395
Title: Genomic and Psychosocial Effects of the Relaxation Response Resiliency Program (3RP) on Patients With MGUS and Smoldering Multiple Myeloma
Brief Title: Genomic and Psychosocial Effects of the 3RP on Patients With MGUS and Smoldering Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-266
Record Dates: First submitted 2013-09-23; First posted 2013-10-07 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
Keywords: Relaxation Response Resiliency Program (3RP); monoclonal gammopathy of undetermined significance; smoldering multiple myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Group (Active Comparator): If the participant is assigned to the Immediate Group, the participant will immediately receive the Relaxation Response Resiliency Program (3RP) intervention (3 months), followed by 3 months of continuing to practice what the participant learned during the intervention.
  Interventions: Behavioral: Relaxation Response Resiliency Program (3RP)
- Waitlist Group (Active Comparator): If the participant is assigned to the Waitlist Group, the participant will wait for 3 months and then receive the full Relaxation Response Resiliency Program (3RP) intervention (3 months).
  Interventions: Behavioral: Relaxation Response Resiliency Program (3RP)

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program (3RP) — The intervention will consist of one intake with a psychologist (approximately 60 minutes), 8 3RP sessions once a week over the course of 8 weeks (approximately 1 hour and 30 minutes each), and one exit visit (approximately 30 minutes) over the course of 3-months. During the intervention, the participant will be asked to practice what the participant has learned in the intervention by listening to a 20-minute audio CD daily. Additionally, the participant will be asked to keep track of their daily practice by filling out an online or paper log. During the 3RP session, the clinician will address any barriers or problems the participant may be having with the daily practice and help to problem solve them with the participant.

SUMMARY:
This research study is evaluating the effects of a mind body medicine intervention called the Relaxation Response Resiliency Program (3RP) on stress and stress related symptoms in patients with monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM).

This research study is a supportive care trial. This means that the intervention program may improve general well-being and comfort, but is not considered a treatment or "cure" for MGUS or SMM. It is considered an investigational intervention because the investigators are examining the effectiveness of a new program - the 3RP - on reducing stress and stress-related symptoms in patients with MGUS and SMM. Standard management of MGUS and SMM involves regular monitoring without chemotherapy. Mind-body medicine, as defined by the National Institutes of Health, "focuses on the interactions among the brain, mind, body, and behavior, and on the powerful ways in which emotional, mental, social, spiritual, and behavioral factors can directly affect health." The 3RP is a newly designed group therapy program that through a variety of mind body principles and self-care interventions seeks to buffer stress and promote psychological resiliency and physical well-being.

This study will examine the effectiveness of the 3RP in reducing stress and symptoms associated with stress in patients diagnosed with MGUS or SMM. Data from this study will also be used to assess changes in gene expression that result from 3RP intervention, particularly genetic pathways that are known to be dysregulated in MM.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing this consent form, the participant will be asked some questions to find out if the participant can be in the research study:

- A medical history, which includes questions about the participant's physical and mental health, current medications, and any allergies.

If these tests show that the participant are eligible to participate in the research study, the participant will receive the study intervention. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

* After the screening procedures confirm that the participant is eligible to participate in the research study:
* Collections Visit One: After the screening visit confirms that the participant is eligible to participate, the participant will be scheduled for Collections Visit One. At Collections Visit One, the participant will complete:
* A demographic questionnaire: This will include questions about the participant's age, gender and ethnicity.
* A series of questionnaires: These will ask the participant's about their overall wellness and take about 30-45 minutes to complete.
* A small blood sample collection: Trained nursing staff will take about 1.5 tablespoons of blood from a single prick to the participant's arm. This procedure will take about 10-15 minutes. This is to provide samples for research tests that may help the investigator's learn more about how the study treatment affects how the participant's genes are expressed.
* OPTIONAL - Bone marrow, plasma and serum collection: This collection is optional and is described in more detail in Section O. Trained nursing staff will take about 1 tablespoon of bone marrow through a standard bone marrow aspirate procedure. This procedure takes about 20-30 minutes to complete, however most of the time is used to get everything ready (such as preparing the skin) as well as 5-10 minutes reserved for relaxing after the procedure is completed. This is to provide samples for research tests that may help the investigator learn more about how the study treatment affects the participant's disease. (This collection is optional and is described in more detail in section O.)
* Since the effect of the study intervention with other medications may not be known, it is important that the participant tell the research doctor about all prescription and non-prescription drugs, herbal preparations and nutritional supplements that the participant is taking or is planning to take.
* Randomization: In order to measure the effects of the intervention, the participant will be "randomized" into one of the study groups after Collections
* Visit One: Immediate Group or Waitlist Control. The Immediate Group will receive the study intervention within two weeks after the Screening and Collections Visit One procedures. Randomization means that the participant is put into a group by chance. It is like flipping a coin. The participant will have an equal chance of being placed in either group. Both groups will receive the same intervention during the course of the study, but at different time points.
* If the participant is assigned to the Waitlist Control group, Collections Visit One will be followed by 3 months of waiting for the intervention. The participant would then attend Collections Visit Two, followed by the intervention (3 months) and then by Collections Visit Three.
* If the participant is assigned to the Immediate Group, Collections Visit One will be followed by the intervention (3 months). the participant would then attend Collections Visit Two, followed by 3 months of continuing to practice what the participant learned during the intervention, and then by Collections Visit Three.
* After Collections Visit One, the participant will be given a group assignment and a calendar of future study visits indicating the potential date, time and locations of the participant's study visits.
* Study Intervention: The intervention will consist of one intake with a psychologist (approximately 60 minutes), 8 3RP sessions once a week over the course of 8 weeks (approximately 1 hour and 30 minutes each), and one exit visit (approximately 30 minutes) over the course of 3-months. All intervention visits will take place at the Benson-Henry Institute for Mind Body Medicine at Massachusetts General Hospital.
* During the intervention (and follow up period for those in the Immediate Group), the participant will be asked to practice what the participant has learned in the intervention by listening to a 20-minute audio CD daily. Additionally, the participant will be asked to keep track of their daily practice by filling out an online or paper log. During the 3RP session, the clinician will address any barriers or problems the participant may be having with the daily practice and help to problem solve them with the participant.
* Collections Visit Two: This visit will be the same as Collections Visit One.
* Collections Visit Three: During this visit, the participant will complete:
* A series of questionnaires: These will ask about the participant's overall wellness, and will take about 30-45 minutes to complete.
* A small blood sample collection: Trained nursing staff will take about 1.5 tablespoons of blood from a single prick to your arm. This procedure takes about 10-15 minutes. This is to provide samples for research tests that may help the investigators learn more about how the study treatment affects how the participant's genes are expressed.
* The investigators will also collect information regarding any changes in the participants medical history since their last visit.

Research Study Plan:

Immediate Group

* Screening Visit: Week 1
* Collections Visit One: Week 1 or 2
* 3RP Session One: Week 3
* 3RP Session Two: Week 4
* 3RP Session Three: Week 5
* 3RP Session Four: Week 6
* 3RP Session Five: Week 7
* 3RP Session Six: Week 8
* 3RP Session Seven: Week 9
* 3RP Session Eight: Week 10
* Collections Visit Two: Week 11/12
* Follow Up Period (home practice): Weeks 13-21 Collections Visit Three: Week 22-24

Waitlist Control

* Screening Visit: Week 1
* Collections Visit One: Week 1 or 2
* Waiting Period: Weeks 2-10
* Collections Visit Two: Week 11 or 12
* 3RP Session One: Week 13
* 3RP Session Two: Week 14
* 3RP Session Four: Week 15
* 3RP Session Five: Week 16
* 3RP Session Six: Week 17
* 3RP Session Seven: Week 18
* 3RP Session Eight: Week 19
* Collections Visit Three: Week 22, 23, or 24
* Planned Follow-up (Immediate Group Only): The investigator would like to keep track of the participant's home practice and medical condition for 12 weeks after completion of the 3RP intervention. The investigator would like to do this by contacting the participant by e-mail or phone once a month to see how the participant is doing. By Keeping in touch with the participant and checking on their practice and condition every month helps the investigator look at the long-term effects of the research study. At the end of the 12 weeks, the participant will come in for their last study visit - the follow up visit, which is described above.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed high-risk monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM) as defined below in table #.

MGUS

* Serum monoclonal protein level < 3 g/dL but > 1.5g/dl,
* Bone marrow plasma cells < 10%
* Non-IgG MGUS (ie IgA, IgM, IgD MGUS)
* Abnormal serum free light chain ratio (ie ratio of kappt to lambda free light chains < 0.26 or > 1.65)
* Absence of end-organ damage, such as lytic bone lesions, anemia, hypercalcemia, or renal failure, that can be attributed to a plasma cell proliferative disorder

SMM (also referred to as asymptomatic multiple myeloma)

* Serum monoclonal protein (IgG or IgA) level > 3 g/dL,
* and /or bone marrow plasma cells > 10%,
* absence of end-organ damage, such as lytic bone lesions, anemia, hypercalcemia, or renal failure, that can be attributed to a plasma cell proliferative disorder
* Participants must be at least 18 years old. Because no dosing or adverse event data are currently available on the use of RR in participants <18 years of age, children are excluded from this study.
* The effects of RR on the developing human fetus are unknown. For this reason, should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants with concurrent active cancer or active cancer with in the last 5 years are ineligible.
* Participants with serious or unstable illness, as determined by study physicians and clinicians, may be deemed unfit to participate.
* Participants with current bipolar or psychotic disorders with active symptoms or treatment within the last 5 year will be excluded.
* Participants will be excluded if they are currently taking (within the last 6 months) psychoactive medications (e.g. mood stabilizers, antipsychotics), with the exception of hypnotics and antidepressants, which will be permitted.
* Participants may not be receiving any other study agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
NF-κB pathway expression in PBMCs | baseline to 3 months
  The expression of the NF-kB pathway in peripheral blood mononuclear cells will be determined on the basis of cumulative expression of normalized copy number of all the genes in the pathway. The genes for the NF-kB pathway will be obtained from the MSigDB (Molecule Signature Database) 3.0 (Broad Institute).

SECONDARY OUTCOMES:
Expression of the previously-defined RR-signature in PBMCs | baseline to 3 months
  The expression of previously-defined RR-signature in peripheral blood mononuclear cells (PBMCs) will be determined on the basis of cumulative expression of normalized copy number of all the genes in the signature. The genes for the signature are defined in Bhasin et al., PLoSOne, 2013.
Gene expression levels in PBMCs | baseline to 3 months
  Normalized gene expression levels in peripheral blood mononuclear cells using nanostring technology.
PSS-10 score | baseline to 3 months
  Change in the 10-item perceived stress scale score.
Normalized gene expression levels in clonal, CD138+ BMPCs | baseline to 3 months
  Normalized gene expression levels in clonal, CD138+ bone marrow plasma cells (BMPCs) measured using nanostring technology.
Beck Anxiety Inventory score | baseline to 3 months
  Change in the Beck Anxiety Inventory score.
Penn State Worry Questionnaire score | baseline to 3 months
  Change in the Penn State Worry Questionnaire score.
LOT-R score | baseline to 3 months
  Change in the Life Orientation Test-Revised score.
MOCS score | baseline to 3 months
  Change in the Measure of Current Status score.

CONTACTS AND LOCATIONS:
Overall Officials: John Denninger, MD/PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Finkelstein-Fox L, Denninger JW, Walsh LE, Laubach JP, Yee AJ, O'Donnell E, Macklin EA, Gu X, Muzikansky A, Libermann TA, Nicolosi G, Richardson PG, Raje NS, Fricchione GL, Perez GK, Traeger LN, Chad-Friedman E, Park ER. Psychosocial and NF-kappaB Activity Effects of the Stress Management and Resiliency Training: Relaxation Response Resiliency Program (SMART-3RP) on Patients With MGUS and Smoldering Multiple Myeloma: A Randomized Waitlist Control Trial. Psychooncology. 2025 Jul;34(7):e70216. doi: 10.1002/pon.70216. PMID 40681960